CLINICAL TRIAL: NCT06320821
Title: ROBOT-ASSISTED KIDNEY TRANSPLANTATION VERSUS OPEN KIDNEY TRANSPLANTATION: a COMPARISON USING PROPENSITY SCORE MATCHING
Brief Title: RAKT OUTCOME ANALYSIS
Status: Enrolling by invitation | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RAKT Version 1.0
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Kidney Transplantation; Robotic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RAKT: robot-assisted kidney transplant patients
- OKT: open kidney transplant patients

SUMMARY:
The goal of this observational study is to compare outcomes of robot-assisted kidney transplantation and open kidney transplantation. The main questions are

- comprehensively analyze our early experience of robot-assisted kidney transplant patients and compare the results with those of open kidney transplant patients

ELIGIBILITY:
Inclusion Criteria:

* Patients received kidney transplantation in SeoulNUH between Jan 2018 and Jan 2024

Exclusion Criteria:

* patients with multi-organ transplant
* patients with missing operative data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study includes patients received kidney-only transplants between Jan 2018 and Jan 2024 in Seoul National University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-08-21 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
learning curve | transplantation to 6 months post-transplant
  The Shewhart control chart and cumulative sum (CUSUM) analysis were used to evaluate technical outcomes and learning curve of RAKT based on RT, NAT, venous anastomosis and arterial anastomosis times

SECONDARY OUTCOMES:
renal function | transplantation to 6 months post-transplant
  This study will compare estimated glomerular filtration rate and graft survival rate between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided